CLINICAL TRIAL: NCT06199531
Title: A Phase 1/2/3 Open-label, Single Arm, Dose-finding Study to Investigate Long-term Safety, Tolerability and Efficacy of GS-100, an Adeno-associated Virus Serotype 9 (AAV9) Vector-mediated Gene Transfer of Human NGLY1, in Patients With NGLY1 Deficiency
Brief Title: Safety and Efficacy of GS-100 Gene Therapy in Patients With NGLY1 Deficiency
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grace Science, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-100-A301
Record Dates: First submitted 2023-11-21; First posted 2024-01-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: NGLY1 Deficiency
Keywords: Gene Therapy; Intervention study; Infusions, Intraventricular; Biomarker; Enzyme Replacement Therapy
MeSH Terms: conditions — NGLY1 deficiency | interventions — d-limonene-medium-chain monoglyceride

STUDY DESIGN:
Intervention Model Description: Dose escalation cohort study of GS-100 administered by intracerebroventricular (ICV) infusion; dose cohorts will be assigned in sequential order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1a (Experimental): 13-18 years old, then 6-12 years old (Low dose GS-100)
  Interventions: Genetic: GS-100
- Cohort 2a (Experimental): 13-18 years old, then 2-5 years old (Mid dose GS-100)
  Interventions: Genetic: GS-100
- Cohort 3a (Experimental): 6-18 years old, then 2-18 years old (High dose GS-100)
  Interventions: Genetic: GS-100

INTERVENTIONS:
Genetic: GS-100 — A single intracerebroventricular (ICV) dose of the study treatment will be administered to patients with confirmed mutations in the NGLY1 gene.
  Other Names: Recombinant, single-stranded adeno-associated virus serotype 9 (AAV9) vector that encodes a full-length version of human NGLY1

SUMMARY:
A non-randomized, open-label, dose escalation study of a single intracerebroventricular (ICV) administration of a gene replacement therapy in subjects who are 2 to 18 years old with NGLY1 Deficiency.

DETAILED DESCRIPTION:
This study is a first in human (FIH) open-label, dose escalation study designed to assess the safety and efficacy of administration of an adeno-associated viral vector serotype 9 (AAV9) carrying the gene encoding N-glycanase 1 (NGLY1) in subjects with NGLY1 Deficiency. The study treatment will be delivered via intracerebroventricular (ICV) injection. All outcomes (primary, secondary, exploratory) will be assessed at 52 weeks. Safety will be monitored continuously throughout the study for adverse / serious adverse events and dose limiting toxicities. Efficacy outcomes will be assessed at baseline and 52 weeks. The co-primary outcomes will be change from baseline in cerebrospinal fluid (CSF) GlcNAc-Asn (GNA, or N-acetylglucosamine), the NGLY1 Deficiency biomarker, and change in motor subdomain on the Bayley Scales of Infant and Toddler Development (BSID-4). Secondary outcomes will include weight (Z-score), clinical and caregiver impressions of change, and other neurocognitive assessment tools. Exploratory outcomes will include brain volumes as measured by magnetic resonance imaging (MRI), quality of life assessments (including sleep habits), liver function test results, and lacrimation assessments. Each participant will be followed for safety and efficacy for 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 2 to 18 years of age, inclusive, at the time of signing the informed consent form (ICF)
* Patients with a documented diagnosis of NGLY1 Deficiency based on detection of biallelic variants in the NGLY1 gene via molecular genetic sequencing
* Elevated GNA levels may be considered alongside genetic sequencing data and other clinical data to assist with diagnosis confirmation
* Patients with two or more of the following clinical features typical of NGLY1 Deficiency:

  1. Global developmental delay and/or intellectual disability
  2. Hyperkinetic movement disorder
  3. Transient elevation of transaminases
  4. (Hypo)alacrima
  5. Peripheral neuropathy
* For patients with epilepsy who require anti-seizure medications for seizure control: must be on a stable regimen for 28 days prior to enrollment
* Patients willing and capable per investigator opinion to comply with study procedures and requirements
* Females of childbearing potential must have a negative serum pregnancy test at screening and must agree to use an acceptable method of highly effective contraception from screening through the end of the study
* Patients or parent(s)/guardian(s) must be willing and able to provide written consent after the nature of the study has been explained and prior to performance of any research-related procedures

Exclusion Criteria:

* Patients at Level 5 of both the Gross Motor Function Classification System Expanded and Revised (GMFCS E&R) and the Communication Function Classification System (CFCS) scales as assessed by the investigator
* Contraindication to use of corticosteroids or history of a condition that could worsen with corticosteroid therapy, as assessed, and determined by the investigator
* Signs / symptoms of increased intracranial pressure (ICP), history of space occupying lesion, or ventricular shunt that would preclude ICV procedures or safety assessments

  a. If clinical signs or symptoms of increased ICP are present (such as headache, vomiting, altered mental status), an ophthalmology examination will be performed to assess for papilledema and/or venous pulsations
* Any comorbid medical or behavioral condition that, in the opinion of the investigator, may adversely affect the safety and well-being of the participant during the study, interfere with completion of the study procedures or follow-up, or compound interpretation of the study results
* Vital signs outside age-based normative values:

  1. Blood pressure: values > 99th percentile as cited in the National Heart, Lung and Blood Institute (NHLBI) guidelines for blood pressure levels based on subject's age, height and sex (nhlbi.nih.gov/files/docs/guidelines/child_tbl.pdf)
  2. Temperature: evidence of fever such as body temperature (e.g., orally measured) of 38.0°C (100.3°F)
  3. Respiratory rate in breaths per minute: toddler (1-3 years old): 24-40; preschooler (4-5 years old): 22-34 breaths per minute; school-aged child (6-12 years old): 18-30 breaths per minute; adolescence (13-18 years old): 12-16.
  4. Oxygen saturation on room air < 92%
* Any condition that in the opinion of the investigator or the study medical monitor would prevent the patient from fully complying with the requirements of the study (including the corticosteroid treatment outline in the protocol) and/or would impact or interfere with the evaluation and interpretation of patient safety or efficacy results
* Known allergy or hypersensitivity to the GS-100 investigational product formulation
* Prior treatment with gene therapy
* Treatment with any investigational product (IP) within 30 days or 5 half-lives of the IP, whichever is longer, prior to screening period. For patients who have received a prior investigational product, all ongoing AEs experienced while receiving the investigational product must have been resolved prior to screening for this study
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study that does not interfere with the requirements of the current protocol and does not have the potential to impact the evaluation of safety and efficacy of GS-100
* Coagulation dysfunction at screening as defined by the following:

  a. INR: ≥1.4 x Upper Limit of Normal (ULN)
* Any current infection with hepatitis B virus (HBV) as evidenced by as evidenced by positive HBV surface antigen (HBsAg), and/or HBV core antibody (HBcAb) at screening. Isolated HBsAb positivity for HBV vaccination in conjunction with negative confirmatory HBV DNA testing at screening is not exclusionary
* Any prior or current infection with hepatitis C virus (HCV) as evidenced by positive HCV antibody testing and confirmed by positive polymerase chain reaction (PCR) RNA testing at screening
* Any of the following abnormal laboratory values:

  1. Hemoglobin level: < 9 g/dL
  2. Absolute neutrophil count: < 1000 cells/microliter
  3. Platelet count: < 100,000/mm3
  4. Creatinine: > 1.25 x ULN
* Have a major surgery planned during the screening period through 52 weeks following GS-100 infusion, including major dental procedures (e.g., wisdom tooth extraction)
* Pregnant or breastfeeding female patient
* Patients that demonstrate elevated serum adrenocorticotropic hormone (ACTH) 1.5 times the upper limit of normal for the reference range must be referred for consultation with a pediatric endocrinologist to rule out primary adrenal insufficiency prior to being enrolled into the study. Patients may re-screen for participation in the study after medical consultation and / or possible treatment has been initiated to address any adrenal insufficiency

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious AEs (SAEs) | 5 years (multiple visits)
Change in liver size by palpation | 5 years (multiple visits)
Complete blood count (CBC) | 5 years (multiple visits)
Coagulation as measured by prothrombin time (PT) | 5 years (multiple visits)
Partial prothrombin time (aPTT) | 5 years (multiple visits)
International normalized ratio (INR) | 5 years (multiple visits)
Gamma-glutamyl transferase (GGT) | 5 years (multiple visits)
Alkaline phosphatase (ALP) | 5 years (multiple visits)
Alanine aminotransferase (ALT) | 5 years (multiple visits)
Serum troponins | 5 years (multiple visits)
Change in nerve conduction velocity (NCV) as assessed by nerve conduction studies | 5 years (multiple visits)
To assess for inflammation or evidence of microgliosis or astrocytosis on MRI | 5 years (multiple visits)
Change in cardiac size as assessed by chamber size and wall thickness on echocardiogram | 5 years (multiple visits)
Change in cardiac function as assessed by ejection fraction on echocardiogram | 5 years (multiple visits)
Sodium (meq/L) | 5 years (multiple visits)
Potassium (meq/L) | 5 years (multiple visits)
Chloride (meq/L) | 5 years (multiple visits)
Bicarbonate (meq/L) | 5 years (multiple visits)
Blood urea nitrogen (BUN) (mg/dL) | 5 years (multiple visits)
Creatinine (mg/dL) | 5 years (multiple visits)
Glucose (mg/dL) | 5 years (multiple visits)
Total protein (g/dL) | 5 years (multiple visits)
Albumin (g/dL) | 5 years (multiple visits)
Total bilirubin (mg/dL) | 5 years (multiple visits)
Direct bilirubin (mg/dL) | 5 years (multiple visits)
Calcium (mg/dL) | 5 years (multiple visits)
Phosphate (mg/dL) | 5 years (multiple visits)
Alkaline phosphatase (U/L) | 5 years (multiple visits)
Lactic dehydrogenase (U/L) | 5 years (multiple visits)

SECONDARY OUTCOMES:
Change from baseline of GNA (GlcNAc-Asn, or N-acetylglucosamine) level in CSF | 5 years (multiple visits)
Change from baseline at 52 weeks in weight (Z-score) | 52 weeks
Change from baseline at 52 weeks in Pediatric Quality of Life Inventory (PedsQL) | 52 weeks
  Total score 0-100; a higher score reflects a higher quality of life
Change from baseline at 52 weeks in Clinical Global Impression of Change (CGI-C) | 52 weeks
  Range from 1-7, with 1 being marked improvement
Change from baseline at 52 weeks in Clinical Global Impression of Severity (CGI-S) | 52 weeks
  Range from 1-7, with 1 being normal/no impairment
Change from baseline at 52 weeks in Caregiver Global Impression of Severity (CaGI-S) | 52 weeks
  Range from 1-7, with 1 being normal/no impairment
Change from baseline at 52 weeks in peripheral nerve function measured by nerve conduction velocity (NCV) in msecs | 52 weeks
Assessment of NGLY1 and capsid-specific cellular immunity by enzyme-linked immunosorbent spot (ELISpot) on peripheral blood mononuclear cells (PBMC) | 5 years (multiple visits)
Detection of antibodies against AAV9 capsid (AAV9 Total antibodies, AAV9 Neutralizing antibodies) and NGLY1 (NGLY1 Total antibodies) | 5 years (multiple visits)
Change from baseline at 52 weeks in Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) | 52 weeks
  Standard scores are based on a mean of 100 and a standard deviation of 15; a higher score reflects a higher level of skill
Change from baseline at 52 weeks in Vineland Adaptive Behavior Scales-3 assessment (Vineland-3) for the Communication, Daily Living skills, Socialization, and Motor domains | 52 weeks
  Standard scores for domains are based on a mean of 100 and a standard deviation of 15; a higher score reflects a higher level of skill
Change from baseline at 52 weeks in Bayley Scales of Infant and Toddler Development 4th Ed (BSID-4) for the Cognitive, Language, and Motor scales | 52 weeks
  Total Raw Scores, Growth Score Values (GSVs), and Age Equivalent Scores will be analyzed; Raw Scores range 0-162; GSVs range 428-559; Age Equivalent Scores range 1-42 months; a higher score reflects a higher level of skill.
Change from baseline at 52 weeks in Gross Motor Function Measure (GMFM) | 52 weeks
  Scores range from 0-264; a higher score reflects a higher level of skill.
Change from baseline at 52 weeks in seizure frequency in subjects with seizures | 52 weeks
Change from baseline at 52 weeks in sitting/standing assessment at 52 weeks | 52 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Oakland Children's Hospital (UCSF Benioff), Oakland, California
  - Columbia University Irving Medical Center, New York, New York
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tong S, Ventola P, Frater CH, Klotz J, Phillips JM, Muppidi S, Dwight SS, Mueller WF, Beahm BJ, Wilsey M, Lee KJ. NGLY1 deficiency: a prospective natural history study. Hum Mol Genet. 2023 Sep 5;32(18):2787-2796. doi: 10.1093/hmg/ddad106. PMID 37379343
- [Background] Stanclift CR, Dwight SS, Lee K, Eijkenboom QL, Wilsey M, Wilsey K, Kobayashi ES, Tong S, Bainbridge MN. NGLY1 deficiency: estimated incidence, clinical features, and genotypic spectrum from the NGLY1 Registry. Orphanet J Rare Dis. 2022 Dec 17;17(1):440. doi: 10.1186/s13023-022-02592-3. PMID 36528660
- [Background] Levy RJ, Frater CH, Gallentine WB, Phillips JM, Ruzhnikov MR. Delineating the epilepsy phenotype of NGLY1 deficiency. J Inherit Metab Dis. 2022 May;45(3):571-583. doi: 10.1002/jimd.12494. Epub 2022 Mar 11. PMID 35243670